CLINICAL TRIAL: NCT02469194
Title: Mechanisms and Predictors of Unusual Radiation or Chemotherapy Toxicity
Status: Withdrawn | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 09915
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Severe or Mild Toxicity From Radiotherapy and/or Chemotherapy
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5-10 cc of whole blood will be obtained using standard, sterile venipuncture techniques
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Blood Draw — 5-10 cc of whole blood will be obtained using standard, sterile venipuncture techniques

SUMMARY:
In general, the toxicity of radiation therapy and chemotherapy exhibits a strong dose-response relationship. However, patients receiving similar doses still exhibit a range of toxicity responses due to a variety of factors, including comorbid conditions, disease (cancer) specific factors, and inter-individual genetic variation. A very small percentage of patients experience side effects that are either extremely severe or extremely mild compared to the majority of patients for the dose of radiation or chemotherapy given. Currently, the reasons for this are not entirely clear, but likely relate to patient specific factors such as immune response, cell/tissue repair capacity and other factors that fundamentally rely on rare genetic variations at loci involved in these responses. For example, patients with homozygous deletions in DNA damage response genes such as ATM are uniquely sensitive to DNA damaging agents. Many patients with severe, homozygous mutations in such genes have other sequela that lead to medical recognition of the syndrome prior to therapy. The investigators hypothesize that patients with unusually severe toxicity from therapy that do not exhibit classical signs of homozygous mutation syndromes are heterozygous for nonfunctional or hypofunctional alleles at these loci, such that the defect is only uncovered under the relatively acute, severe stress on that pathway by radiation or chemotherapy. Conversely, patients with very mild reactions could exhibit rare variants/combinations of variants that make them uniquely resistant to chemotherapy or radiotherapy toxicity.

The purpose of the study is to better understand these mechanisms with the eventual goal of developing predictive markers that will allow us to help individually tailor cancer therapy is in future patients. Will accomplish these goals by studying a variety of factors from a single vial of blood. These will include circulating proteins and hormones, circulating cells and the levels and sequences of white blood cell DNA or RNA using a variety of techniques including but not limited to determination of cytokine/hormone levels, proteomic analysis, immunocytochemical assays, whole exome sequencing and qPCR.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be age 18 or greater Subjects will have undergone chemotherapy and/or radiotherapy and experienced unusually mild or severe toxicity.

Exclusion Criteria:

* Subjects for who, after initial review of medical records by study team personnel are not judged by the PI and/or sub-investigators to have sufficiently unusual toxicity from therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the inpatient and outpatient clinical practices in the University of Pennsylvania Health System. There will be no attempt to advertise enrollment on this protocol to physicians outside of the treating departments (i.e. Radiation Oncology, Surgery, Medical Oncology).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Keith Cengel, MD, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States